CLINICAL TRIAL: NCT04217967
Title: A Multicenter, Open-label, Prospective Study of Ixazomib, Lenalidomide, and Ixazomib in Combination With Lenalidomide for Maintenance Therapy in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Ixazomib, Lenalidomide, and Combination for Maintenance in NDMM Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Beijing Jishuitan Hospital (Other); Beijing Chao Yang Hospital (Other); Xuanwu Hospital, Beijing (Other); Peking University First Hospital (Other); Jilin Provincial Tumor Hospital (Other); Second Hospital of Shanxi Medical University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Tianjin Medical University General Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Shanxi Bethune Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Junling Zhuang, Professor, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-2129
Record Dates: First submitted 2020-01-01; First posted 2020-01-06 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: real-world; dual-drug maintenance; oral regimen
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lenalidomide group (Active Comparator): lenalidomide 25mg qod d1~21 days, rest 7 days
  Interventions: Drug: Lenalidomide
- Ixazomib group (Active Comparator): ixazomib 4mg orally, once a week, 3 times a month
  Interventions: Drug: Ixazomib
- Combination group (Experimental): ixazomib 4mg orally, once a week, 3 times a month lenalidomide 25mg qod d1~21 days, rest 7 days use in combination
  Interventions: Drug: Ixazomib; Drug: Lenalidomide

INTERVENTIONS:
Drug: Ixazomib — the ixazomib group uses ixazomib as the comparator group, the combination group receives both lenalidomide and ixazomib as the experimental group
  Arms: Combination group; Ixazomib group
Drug: Lenalidomide — the lenalidomide group uses lenalidomide as comparitor group and the combination group receives both lenalidomide and ixazomib
  Arms: Combination group; Lenalidomide group

SUMMARY:
The purpose of this study is to evaluate the real-world efficacy and safety of ixazomib, lenalidomide, or ixazomib in combination with lenalidomide as maintenance therapy in patients with newly diagnosed multiple myeloma in China.

DETAILED DESCRIPTION:
Multiple myeloma (MM), the second most common hematological malignancy, is a clonal plasma cell disorder characterized by the secretion of monoclonal immunoglobulins. The annual incidence of newly diagnosed MM (NDMM) patients is about 2-3/100,000. In the past 20 years, the median overall survival (OS) of MM patients has prolonged from 3 to 5 years to 8 to 10 years since many novel agents developed on the pipeline of treatment. Moreover, multi-drug combination chemotherapy, low-intensity maintenance therapy after achieving a certain effect also contributed to improving the progression-free survival (PFS) and OS in MM patients. Therefore, many international guidelines have explicitly recommended maintenance therapy after first-line regimens until disease progression.

Common maintenance medications include immunomodulatory drugs (IMiDs) such as lenalidomide, thalidomide, ect; proteasome inhibitors (PIs) such as bortezomib. Among them, lenalidomide has the most reliable data as maintenance therapy for prolonging PFS. Although bortezomib maintenance has shown advantages in high-risk MM patients in some clinical trials, it has poor compliance in the real world due to the injection mode of administration and peripheral neuropathy (PN) after long-term use. There is currently no data on the maintenance of large-scale cases in China. The maintenance of regimens in the real world is not standardized, including drug dosage and duration of application. In addition, due to the high cost of bortezomib or lenalidomide for long-term application, domestic thalidomide still accounts for a certain proportion, but its side effects especially PN are very prominent. In addition to the proven efficacy, MM maintenance treatments should preferably include good tolerability, manageable toxicities and administration convenience.

The second-generation PI drug, Ixazomib, was approved in China in May 2018. Based on the data of TOURMALINE MM1 trial and China extended study, ixazomib was approved for the treatment of relapsed and refractory MM. Further more, recent maintenance study after autologous transplantation (MM3) suggested that ixazomib significantly prolonged PFS for 6 months compared with placebo. Because ixazomib is an oral form with a few side effects, especially less PN than bortezomib, safety data and compliance of ixazomib in the real world were comparable as those in the clinical trials.

The survival of patients with multiple myeloma in China is worse than that of western countries. One of the important reasons is irregular follow-up and nonstandard maintenance therapies. Many Chinese MM patients still use traditional maintenance drug thalidomide, which is difficult to apply for a long time due to toxicities especially PN and gastrointestinal reactions. The second generation IMiD drug lenalidomide as maintenance treatment has been increasingly accepted by patients and hematologists. However, due to the low proportion of autologous stem cell transplantation (ASCT) after first-line regimens in China, the efficacy of single-agent maintenance is also limited, especially for high-risk patients. As novel anti-myeloma drugs were rapidly approved and reimbursed in China, a dual oral maintenance regimen of lenalidomide in combination with ixazomib is being explored.

The purpose of this multi-centered study is to evaluate the real world efficacy and safety of the maintenance therapies in Chinese patients with newly diagnosed multiple myeloma (NDMM), non-transplant; which include ixazomib monotherapy, ixazomib combined with lenalidomide, and lenalidomide monotherapy.

Adult NDMM patients who acquire at least partial response (PR) after 4~9 cycles of front-line regimens including ASCT will be recruited. Those who do not reach a PR after 4 cycles of front-line regimens will be switched to the second regimen for at most 5 cycles. After reaching a PR, these patients will also be recruited to the study. Maintenance therapies will be classified into three groups depending on patients' and doctors' discretion, including ixazomib 4mg day 1, 8,15; lenalidomide 25mg qod day 1~21; ixazomib and lenalidomide combination with same doses. Front-line maintenance is given till disease progression. Progression free survival and safety issues will be recorded. Drug doses will be adjusted or withdrawn based on the degree of toxicities.

Adjunctive treatments are prophylaxis of herpes zosters with acyclovir, prophylaxis of venous thrombotic events with aspirin, prophylaxis of high-risk infections with sulfanilamide. The doses of lenalidomide are adjusted depending on clearance of creatinine.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 18 years;
2. Newly diagnosed MM patients who fulfill the diagnostic criteria of International Myeloma Working Group (IMWG) 2014 standard; transplant-ineligible or transplant eligible yet without intent for ASCT
3. Maintenance treatment will start after first-line treatment or second-line treatment;
4. The total courses of front-line regimens are between 4-9;
5. The clinical efficacy before the enrollment is partial response (PR) or better;
6. Physical performance status (ECOG) score ≤ 2;
7. Patients participate in the study based on his/her own will and voluntarily sign the informed consent form

Exclusion Criteria:

1. Patients who are allergic or intolerant to ixazomib or lenalidomide;
2. patients with severe cardiopulmonary dysfunction;
3. patients with severe hepatic insufficiency, ALT or bilirubin more than 2 times the upper limits of normal range;
4. patients with other malignancies (except for carcinoma in situ);
5. patients with serious bacterial or viral infections, such as HIV or HBV, HCV, etc.;
6. pregnant or lactating women;
7. can not be strictly contraceptive;
8. Psychiatric patients and patients with other serious mental illness that potentially impact signing informed consent and disease consultation and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
progression-free survival | From date of enrollment until the date of first documented progression, assessed up to 20 months
  from enrollment to first disease progression
overall survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  from enrollment to death with follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Junling Zhuang, MD, Principal Investigator — Peking Union Medical College, department of hematology
Locations (1):
- PekingUMCH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
individual baseline characteristic, treatment and follow-up results will be shared after publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication, the data will become available

REFERENCES:
- [Background] Palumbo A, Anderson K. Multiple myeloma. N Engl J Med. 2011 Mar 17;364(11):1046-60. doi: 10.1056/NEJMra1011442. No abstract available. PMID 21410373
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Anderson KC. Progress and Paradigms in Multiple Myeloma. Clin Cancer Res. 2016 Nov 15;22(22):5419-5427. doi: 10.1158/1078-0432.CCR-16-0625. PMID 28151709
- [Background] Gay F, Jackson G, Rosinol L, Holstein SA, Moreau P, Spada S, Davies F, Lahuerta JJ, Leleu X, Bringhen S, Evangelista A, Hulin C, Panzani U, Cairns DA, Di Raimondo F, Macro M, Liberati AM, Pawlyn C, Offidani M, Spencer A, Hajek R, Terpos E, Morgan GJ, Blade J, Sonneveld P, San-Miguel J, McCarthy PL, Ludwig H, Boccadoro M, Mateos MV, Attal M. Maintenance Treatment and Survival in Patients With Myeloma: A Systematic Review and Network Meta-analysis. JAMA Oncol. 2018 Oct 1;4(10):1389-1397. doi: 10.1001/jamaoncol.2018.2961. PMID 30098165
- [Background] Dimopoulos MA, Gay F, Schjesvold F, Beksac M, Hajek R, Weisel KC, Goldschmidt H, Maisnar V, Moreau P, Min CK, Pluta A, Chng WJ, Kaiser M, Zweegman S, Mateos MV, Spencer A, Iida S, Morgan G, Suryanarayan K, Teng Z, Skacel T, Palumbo A, Dash AB, Gupta N, Labotka R, Rajkumar SV; TOURMALINE-MM3 study group. Oral ixazomib maintenance following autologous stem cell transplantation (TOURMALINE-MM3): a double-blind, randomised, placebo-controlled phase 3 trial. Lancet. 2019 Jan 19;393(10168):253-264. doi: 10.1016/S0140-6736(18)33003-4. Epub 2018 Dec 10. PMID 30545780
- [Background] Chakraborty R, Muchtar E, Kumar SK, Buadi FK, Dingli D, Dispenzieri A, Hayman SR, Hogan WJ, Kapoor P, Lacy MQ, Leung N, Warsame R, Kourelis T, Gonsalves W, Gertz MA. Outcomes of maintenance therapy with lenalidomide or bortezomib in multiple myeloma in the setting of early autologous stem cell transplantation. Leukemia. 2018 Mar;32(3):712-718. doi: 10.1038/leu.2017.256. Epub 2017 Aug 14. PMID 28848227
- [Background] Kumar SK, Berdeja JG, Niesvizky R, Lonial S, Laubach JP, Hamadani M, Stewart AK, Hari P, Roy V, Vescio R, Kaufman JL, Berg D, Liao E, Rajkumar SV, Richardson PG. Ixazomib, lenalidomide, and dexamethasone in patients with newly diagnosed multiple myeloma: long-term follow-up including ixazomib maintenance. Leukemia. 2019 Jul;33(7):1736-1746. doi: 10.1038/s41375-019-0384-1. Epub 2019 Jan 29. PMID 30696949